CLINICAL TRIAL: NCT02889523
Title: A Phase Ib-II Study of Tazemetostat (EPZ-6438) in Newly Diagnosed Diffuse Large B Cell Lymphoma (DLBCL) or High Risk Follicular Lymphoma (FL) Patients Treated by R-CHOP
Brief Title: Study of Tazemetostat in Newly Diagnosed Diffuse Large B Cell and Follicular Lymphoma Patients Treated by Chemiotherapy
Acronym: Epi-RCHOP
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Epizyme, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Epi-RCHOP
Record Dates: First submitted 2016-07-11; First posted 2016-09-05 (Estimated); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Lymphoma; DLBCL; Follicular Lymphoma
Keywords: Front line therapy; Age-adjusted International Prognostic Index (aa-IPI) >1; 60 to 80 years
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — tazemetostat; Rituximab; Cyclophosphamide; Vincristine; Doxorubicin; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DLBCL cohort (Experimental): RCHOP + tazemetostat:
  - RCHOP: rituximab (IV, 375 mg/m², day 1), Prednisolone (PO, 40 mg/m² in the morning, day 1 to day 5), doxorubicine (IV, 50 mg/m², day 1), cyclophosphamide (IV, 750 mg/m², day 1), vincristine (IV, 1.4 mg/m², day 1): Phase I : 8 cycles, every 21 days Phase II : 6 cycles, every 21 days
  * Rituximab (IV, 375 mg/m², day 1) Phase II : 2 cycles, every 21 days
  * Tazemetostat: PO, doses according to dose cohorts for phase I, and at RP2D for phase II: continuous: Cycle 1: 2 to 21 BID, Cycle 2-8: 1 to 21 BID
  Interventions: Drug: Tazemetostat; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin; Drug: Prednisolone
- FL cohort (Experimental): RCHOP + tazemetostat:
  Induction
  * RCHOP: rituximab (IV, 375 mg/m², day 1), Prednisolone (PO, 40 mg/m² in the morning, day 1 to day 5), doxorubicine (IV, 50 mg/m², day 1), cyclophosphamide (IV, 750 mg/m², day 1), vincristine (IV, 1.4 mg/m², day 1):
    6 cycles, every 21 days
  * Rituximab (IV, 375 mg/m², day 1) Phase II : 2 cycles, every 21 days
  * Tazemetostat: PO, RP2D, continuous: Cycle 1: 2 to 21 BID, Cycle 2-8: 1 to 21 BID
  Maintenance
  * Tazemetostat : 6 months (every 8 weeks)
  * Rituximab : 24 months (every 8 weeks)
  Interventions: Drug: Tazemetostat; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin; Drug: Prednisolone

INTERVENTIONS:
Drug: Tazemetostat — Tablets 200 mg, to be administrated per os
  Other Names: EPZ-6438
Drug: Rituximab — 375 mg/m²/dose, D1
  Other Names: Mabthera
Drug: Cyclophosphamide — 750 mg/m²/dose, D1
Drug: Vincristine — 1.4 mg/m²/dose (max 2 mg), D1
Drug: Doxorubicin — 50 mg/m²/dose, D1
Drug: Prednisolone — 40 mg/m2 in the morning D1 to D5

SUMMARY:
Phase I of the study is designed to determine the recommended phase II dose (RP2D) for tazemetostat in patients treated with 8 cycles of R-CHOP 21.

Phase II of the study is designed to determine the safety and the efficacy of tazemetostat in DLBCL and FL patients :

DLBCL : tazemetostat with 6 cycles of R-CHOP 21 + 2 cycles of Rituximab FL : tazemetostat with 6 cycles of R-CHOP 21 + 2 cycles of Rituximab then maintenance with 6 months of tazemetostat and 24 months of Rituximab

DETAILED DESCRIPTION:
Phase I:

Up to 18 patients will be recruited, using a conventional dose-escalation algorithm (3+3 patients per dose level) to identify the maximum tolerated dose (MTD) which will be deemed the RP2D. Patients will receive 8 cycles of RCHOP every 21 days and tazemetostat every day, starting on day 2 of cycle 1.

4 cohorts are defined, according to dose levels of tazemetostat: 400mg Twice a day (BID) (cohort 1, starting level), 600mg BID (cohort 2), 800mg BID (cohort 3), 200mg BID (cohort -1), depending on the observed toxicities.

Phase II:

Up to 184 patients (122 DLBCL and 62 FL) will be recruited and treated with tazemetostat at the MTD and RCHOP.

Patients will receive 6 cycles of RCHOP every 21 days and tazemetostat at the MTD every day, starting on day 2 of cyle 1, + 2 cycles of Rituximab+tazemetostat. For FL, a maintenance of tazemetostat (6 months) + rituximab (24 months) is expected

ELIGIBILITY:
* INCLUSION CRITERIA

  * for Cohort DLBCL ONLY

    * 1-Patients with an untreated DLBCL de novo or transformed from indolent lymphoma (CD 20 positive) with

      * Phase Ib aaIPI ≥ 2
      * Phase II: aaIPI ≥ 1ONLY
    * 2. Age between 60 and 80 years included
  * for Cohort FOLLICULAR ONLY

    * 1-High Tumor Burden (as defined by GELF criteria > 0) frontline follicular lymphoma (FL) with high risk FLIPI 3-5
    * 2. Aged between 18 years and 80 years included
    * 11bis. Females of childbearing potential (FCBP) must agree to use one reliable form of contraception or to practice complete abstinence from heterosexual contact during the following time periods related to this study: 1) for at least 28 days before starting study drug; 2) while participating in the study; 3) dose interruptions; and 4) for at least 12 months after discontinuation of any study treatments (R-CHOP, tazemetostat, Rituximab)
  * For both Cohorts

    * 1bis- For phase II patients: Bi-dimensionally measurable disease defined by at least one single node or tumor lesion > 1.5 cm assessed by CT scan and/or clinical examination AND a FDG avid disease by PETscan
    * 3.ECOG performance status of 0, 1 or 2 (0 or 1 only for phase Ib)
    * 4.Signed informed consent
    * 5.Life expectancy of ≥ 90 days (3 months) before starting tazemetostat
    * 6.Adequate renal function as calculated by a creatinine clearance > 40 mL/min by local institutional formula
    * 7. Adequate bone marrow function as defined as:

      * ANC ≥ 1500/mm3 (≥ 1.5 X 109/L)
      * Platelets ≥ 75,000/mm3 (≥ 75 X 109/L) without platelet transfusion dependency during the last 7 days
      * Hemoglobin ≥ 9 g/dL (may receive transfusion)
    * 8. Adequate liver function as defined as:

      * Total bilirubin ≤ 1.5 × the upper limit of normal (ULN) except for unconjugated hyperbilirubinemia of Gilbert's syndrome
      * Alkaline phosphatase (in absence of bone disease), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 X ULN (or ≤ 5 X ULN if related to lymphoma involvement)
      * Patients with prior Hepatitis B and C are eligible if, for Hepatitis B detection, surface antigen is negative and/or HBV DNA is undetectable, and for Hepatitis C detection, if HCV RNA is undetectable.
    * 9. Left ventricular ejection fraction (LVEF) ≥ 50% of echocardiography or multiple gated acquisition (MUGA) scan
    * 10. Adequate tissue (surgical excision is recommended) for central pathology review and biological caracterisation (see appendix 11
    * 11. Males with partners of childbearing potential must agree to use reliable forms of contraception during 12 months after last treatment administration
    * 12. Patient covered by any social security system (for France only)
    * 13. Patient who understands and speaks one of the country official languages
* EXCLUSION CRITERIA

  * for Cohort DLBCL

    ___15-Previous treatment for B cell lymphoma, except glucocorticoids (no more than 7 days before inclusion, 1 mg/kg/day max)
  * for Cohort FOLLICULAR ONLY

    * 14bis. Prior therapy for lymphoma including radiotherapy except glucocorticoids (no more than 7 days before inclusion, 1 mg/kg/day max)
    * 17-Pregnant or lactating females
  * For both Cohorts

    * 1-Central nervous system or meningeal involvement
    * 2-Contraindication to any drug contained in the chemotherapy regimen
    * 3-Prior treatment with tazemetostat or other inhibitor of EZH2
    * 4-Patients who are undergoing active treatment for another malignancy, exceptions include: A patient who has been disease free for 2 years, or a patient with a history of a completely resected non-melanoma skin cancer or successfully treated in situ carcinoma is eligible Patients with prior history of myeloid malignancies, including myelodysplastic syndrome (MDS) or Acute Myeloid Leukemia(AML) or prior history of T-LBL/T-ALL are excluded whatever receiving treatment or not and whatever date of diagnosis of these pathologies
    * 5-Patients taking medications that are known potent CYP3A4 inducers/inhibitors (including St. John's wort)
    * 6-Patients unwilling to exclude St. John's wort, Seville oranges, grapefruit juice and/or grapefruit from diet
    * 7-Major surgery within 4 weeks before first dose of study drug (minor procedures including transcutaneous biopsy, central line placement are permitted within 2 weeks of enrollment)
    * 8-Inability to take oral medication or malabsorption syndrome or any other uncontrolled gastrointestinal condition that would impare ability to take tazemetostat
    * 9-Significant cardiovascular impairment: congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months of first dose of tazemetostat or ventricular arrhythmia
    * 10-Not applicable
    * 11-Active uncontrolled infection requiring systemic therapy
    * 12-Congenital immunodeficiency or known HIV (human immunodeficiency virus infection)
    * 13-Any other major illness, that in the investigator's judgement, will substantially increase the risk associated with the patient's participation in the study
    * 14-Patients who have undergone a solid organ transplant
    * 16-Treatment with any investigational drug or device within 30 days before planned first cycle of chemotherapy
    * 18-Person deprived of his/her liberty by a judicial or administrative decision
    * 19-Adult person under legal protection
    * 20-Person hospitalized without consent
    * 21-Adult person unabled to provide informed consent because of intellectual impairment, any serious medical condition, laboratory abnormality or psychiatric illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Phase I : Number of Dose Limiting Toxicities | 1 cycle (1 cycle is 21 days)
  Incidence and severity of treatment-emergent AEs qualifying as protocol defined DLT's in cycle 1 and 2 in order to establish the MTD/RP2D
Phase I : Number of Dose Limiting Toxicities | 2 cycles (1 cycle is 21 days)
  Incidence and severity of treatment-emergent AEs qualifying as protocol defined DLT's in cycle 1 and 2 in order to establish the MTD/RP2D
Phase II - DLBCL Cohort : Complete Response Rate based on local assessment | 8 cycles (1 cycle is 21 days)
  Complete response rate as determined by Cheson International Work Group (IWG) 2014: Lugano Classification (Deauville scale 1-3)
Phase II - FL Cohort : Complete Response Rate based on local assessment | 8 cycles (1 cycle is 21 days)
  Complete response rate as determined by Cheson IWG 2014: Lugano Classification (Deauville scale 1-3)

SECONDARY OUTCOMES:
Phase I : Serum concentration of CHOP components in presence/absence of Tazemetostat | Change between baseline - 1 month
Phase I : Serum concentration of Tazemetostat and its metabolite (EZH 6930) in presence of CHOP | Change between baseline - 1 month
Phase I : Complete response rate (CRR) by central review using Cheson IWG criteria | 8 cycles (1 cycle is 21 days)
Phase II - DLBCL Cohort : Number of Adverse Events (AE)/Serious Adverse Events (SAE) | 8 cycles (1 cycle is 21 days)
Phase II - DLBCL Cohort : Complete response rate (CRR) by central review using Cheson IWG criteria | 8 cycles (1 cycle is 21 days)
Phase II - DLBCL Cohort : Overall response rate (ORR) by central review | 52 weeks
Phase II - DLBCL Cohort : Overall response rate (ORR) by central review | 104 weeks
Phase II - DLBCL Cohort : progression free survival (PFS) | 52 weeks
Phase II - DLBCL Cohort : progression free survival (PFS) | 104 weeks
Phase II - DLBCL Cohort : duration of response (DR) | 52 weeks
Phase II - DLBCL Cohort : duration of response (DR) | 104 weeks
Phase II - DLBCL Cohort : overall survival (OS) | 52 weeks
Phase II - DLBCL Cohort : overall survival (OS) | 104 weeks
Phase II - DLBCL Cohort : best overall response (BOR) | 104 weeks
Phase II - FL cohort : Number of AE/SAE | 8 cycles (1 cycle is 21 days)
Phase II - FL cohort : Number of AE/SAE | 13 months
Phase II - FL cohort : PET Complete Response Rate (PET-CRR) by central review according to Lugano 2014 criteria | 8 cycles (1 cycle is 21 days)
Phase II - FL cohort : Complete Response Rate (CRR) | 31 months
Phase II - FL cohort : Overall Response Rate (CRR) | 31 months
Phase II - FL cohort : Progression Free Survival (PFS) | 24 months
Phase II - FL cohort : Progression Free Survival (PFS) | 31 months
Phase II - FL cohort : Event Free Survival (EFS) | 24 months
Phase II - FL cohort : Overall Survival (OS) | 24 months
Phase II - FL cohort : Duration of Response (DR) | 31 months
Phase II - FL cohort : Best Overall Response | 31 months

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ribrag, MD, Study Chair — Institut Gustave Roussy Cancer Campus Grand Paris; Clémentine Sarkozy, MD, Study Chair — Institut Gustave Roussy Cancer Campus Grand Paris; Franck Morshhauser, Pr, Study Chair — Centre Régional Hospitalier de Lille; Loic Ysebaert, MD, Study Chair — IUCT Oncopole de Toulouse
Locations (31):
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - CHU de Liege, Liège
  - CHRU Mont Godinne, Yvoir
- France (28):
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - CH d'Avignon - Hôpital Henri Dufaut, Avignon
  - CHU de Besançon - Hôpital Jean Minjoz, Besançon
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CH de Chambéry, Chambéry
  - CHU d'Estaing, Clermont-Ferrand
  - APHP - Hopital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CHU Grenoble, Grenoble
  - CH Départemental de Vendée, La Roche-sur-Yon
  - CHRU Lille - Hôpital Claude Huriez, Lille
  - Chu de Limoges - Hopital Dupuytren, Limoges
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmette, Marseille
  - CHU de Montpellier - Hôpital Saint-Eloi, Montpellier
  - CHU de Nantes - Hôtel Dieu, Nantes
  - APHP - Hôpital de la Pitié Salpetrière, Paris
  - APHP - Hôpital Saint Louis, Paris
  - CH de Perpigan, Perpignan
  - CHU Lyon Sud, Pierre-Bénite
  - Chu de Poitiers - Hopital de Miletrie, Poitiers
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Rene Hugenin, Saint-Cloud
  - Institut de cancérologie de la Loire, Saint-Priest-en-Jarez
  - CHRU de Strasbourg, Strasbourg
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarkozy C, Morschhauser F, Dubois S, Molina T, Michot JM, Cullieres-Dartigues P, Suttle B, Karlin L, Le Gouill S, Picquenot JM, Dubois R, Tilly H, Herbaux C, Jardin F, Salles G, Ribrag V. A LYSA Phase Ib Study of Tazemetostat (EPZ-6438) plus R-CHOP in Patients with Newly Diagnosed Diffuse Large B-Cell Lymphoma (DLBCL) with Poor Prognosis Features. Clin Cancer Res. 2020 Jul 1;26(13):3145-3153. doi: 10.1158/1078-0432.CCR-19-3741. Epub 2020 Mar 2. PMID 32122924